CLINICAL TRIAL: NCT04788017
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Sequential Parallel Group, Single Ascending Dose Study Evaluating the Safety, Tolerability, and Pharmacokinetics of Ziresovir in Healthy Subjects
Brief Title: A Study Evaluating the Safety, Tolerability, and Pharmacokinetics of Ziresovir in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Ark Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: AK0529-3001
Record Dates: First submitted 2021-02-01; First posted 2021-03-09 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — ziresovir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ziresovir (Active Comparator): The study drugs will be administered to subjects by CRU staff at approximately 8:00 a.m. (± 1 hour), following an overnight fast.
  Immediately following administration of the assigned dose of the study drugs, subjects will be given water such that their water consumption is approximately 240 mL as follows:
  * If administered 60 mL as the study drug dose, follow with approximately 180 mL water.
  * If administered 120 mL as the study drug dose, follow with approximately 120 mL water.
  * If administered 180 mL as the study drug dose, follow with approximately 60 mL water.
  Interventions: Drug: Ziresovir
- placebo (Placebo Comparator): The study drugs will be administered to subjects by CRU staff at approximately 8:00 a.m. (± 1 hour), following an overnight fast.
  Immediately following administration of the assigned dose of the study drugs, subjects will be given water such that their water consumption is approximately 240 mL as follows:
  * If administered 60 mL as the study drug dose, follow with approximately 180 mL water.
  * If administered 120 mL as the study drug dose, follow with approximately 120 mL water.
  * If administered 180 mL as the study drug dose, follow with approximately 60 mL water.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Ziresovir — Planned treatments are:
  * Cohort 1: 300 mg of ziresovir
  * Cohort 2: up to 600 mg of ziresovir
  * Cohort 3: up to 900 mg of ziresovir
  Other Names: AK0529
  Arms: ziresovir
Other: Placebo — Planned treatments are:
  * Cohort 1: 300 mg of placebo
  * Cohort 2: up to 600 mg of placebo
  * Cohort 3: up to 900 mg of placebo
  Arms: placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, dose escalation study to evaluate the safety, tolerability, and pharmacokinetics (PK) of ziresovir following a single ascending oral dose administration in healthy adult subjects under fasted conditions.

DETAILED DESCRIPTION:
Up to 3 dose cohorts are planned. The ziresovir dose level of each cohort is determined based on the collective clinical and nonclinical data of ziresovir.

The proposed dose levels of Cohorts 1, 2 and 3 are 300 mg and up to 600 mg and up to 900 mg, respectively.

A total of up to 24 subjects will be randomized with 18 subjects to receive active drug and 6 subjects to receive placebo in a double-blind fashion. Eight subjects will be randomized in each dose cohort, with 6 subjects to receive active drug and 2 subjects o receive placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of giving written informed consent and complying with study procedures;
2. Between the ages of 18 and 55 years, inclusive;
3. Body mass index (BMI) of 18.0 to 32.0 kg/m2 inclusive and body weight not less than 50 kg;
4. Female subjects must have a negative pregnancy test result at screening;
5. Considered healthy by the Investigator, based on subject's reported medical history, full physical examination, 12-lead ECG, and vital signs;
6. Willing and being able to adhere to study restrictions and to be confined at the Clinical Research Unit.

Exclusion Criteria:

1. Clinically significant reported history of gastrointestinal, cardiovascular, musculoskeletal, endocrine, hematologic, psychiatric, renal, hepatic, bronchopulmonary, neurologic, immunologic, lipid metabolism disorders, or drug hypersensitivity as determined by the Investigator;
2. Poor venous access;
3. Taken an investigational drug or participated in a clinical trial evaluating an investigational drug or device within 30 days (or 5 half-lives) prior to the study drug dose, whichever is longer;
4. Taken any prescription medications within 14 days or 5 half-lives (whichever is longer) of the study drug dose;
5. Major surgery or hospitalization within 6 months prior to screening that in the Investigator's opinion would put the subject or study conduct at risk, or have any scheduled surgery or hospitalization during the study period;
6. Any condition or finding that in the Investigator's opinion would put the subject or study conduct at risk if the subject were to participate in the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2021-03-24 (Actual); Primary Completion 2021-06-14 (Actual); Study Completion 2021-07-22 (Actual)

PRIMARY OUTCOMES:
numbers of all AEs | through study completion, an average of 22 days
  The Common Terminology Criteria for Adverse Events (CTCAE) Version 5 will be used to grade AEs
percentages of all AEs | through study completion, an average of 22 days
  The Common Terminology Criteria for Adverse Events (CTCAE) Version 5 will be used to grade AEs
change from baseline in systolic and diastolic blood pressure | screen/day -1/day 1/day 2/day 3/day4
  blood pressure in millimeter of mercury
change from baseline in pulse rate | screen/day -1/day 1/day 2/day 3/day4
  pulse rate in times per minute
change from baseline in respiratory rate | screen/day -1/day 1/day 2/day 3/day4
  respiratory rate in times per minute
change from baseline in oral temperature | screen/day -1/day 1/day 2/day 3/day4
  oral temperature in degree
change from baseline in Prothrombin time/International Normalized Ratio | screen/day -1/day 2/day4
  INR is calculated from the PT and allows for worldwide standardization of results.
change from baseline in Thrombin time | screen/day -1/day 2/day4
  Thrombin time in seconds
change from baseline in activated Partial Thromboplastin time | screen/day -1/day 2/day4
  activated Partial Thromboplastin time in seconds
change from baseline in Hemoglobin (Hgb) count | screen/day -1/day 2/day4
  Hemoglobin (Hgb) in gram per liter
change from baseline in Hematocrit (Hct) | screen/day -1/day 2/day4
change from baseline in Platelet count | screen/day -1/day 2/day4
  Platelet count per liter
change from baseline in Red blood cell (RBC) count | screen/day -1/day 2/day4
change from baseline in White blood cell (WBC) count with differential | screen/day -1/day 2/day4
change from baseline in Specific gravity from urinalysis | screen/day -1/day 2/day4
change from baseline in pH from urinalysis | screen/day -1/day 2/day4
change from baseline in Protein from urinalysis | screen/day -1/day 2/day4
change from baseline in Glucose from urinalysis | screen/day -1/day 2/day4
change from baseline in Ketones from urinalysis | screen/day -1/day 2/day4
change from baseline in Bilirubin from urinalysis | screen/day -1/day 2/day4
change from baseline in Blood from urinalysis | screen/day -1/day 2/day4
change from baseline in Nitrites from urinalysis | screen/day -1/day 2/day4
change from baseline in Leukocytes from urinalysis | screen/day -1/day 2/day4
change from baseline in Urobilinogen from urinalysis | screen/day -1/day 2/day4
Incidence of abnormal Microscopic urine analysis | screen/day -1/day 2/day4
change from baseline in heart rate-corrected QT interval from resting 12-lead ECGs | screen/day -1/day1/day2/day4
  ECGs will be performed after the subject has been supine for at least 5 minutes
change from baseline in heart rate from resting 12-lead ECGs | screen/day -1/day1/day2/day4
  ECGs will be performed after the subject has been supine for at least 5 minutes
change from baseline in QRS intervals from resting 12-lead ECGs | screen/day -1/day1/day2/day4
  ECGs will be performed after the subject has been supine for at least 5 minutes
change from baseline in treatment-emergent T-wave morphology from resting 12-lead ECGs | screen/day -1/day1/day2/day4
  ECGs will be performed after the subject has been supine for at least 5 minutes
change from baseline in appearance of U-waves from resting 12-lead ECGs | screen/day -1/day1/day2/day4
  ECGs will be performed after the subject has been supine for at least 5 minutes
Incidence of abnormal physical findings | screen/day -1/day2/day3/day4
  full physical examination will be conducted at screening and an abbreviated physical exam will be conducted on Day -1 and Day 2. A symptom-directed physical exam will be conducted on Day 3 and Day 4.

SECONDARY OUTCOMES:
To characterize the drug concentration of ziresovir following single ascending doses by oral administration in healthy adult male and female subjects | 0 (within 90 minutes prior to dosing) and 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48, and 72 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Jimmy Gu, Study Director — Ark Biosciences
Locations (1):
- Frontage, Secaucus, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No